CLINICAL TRIAL: NCT06143644
Title: The Predictive Value of Postoperative Circulating Tumor DNA Monitoring in Assessing the Risk of Recurrence in Stage I-IV Colorectal Cancer Patients, An Observational Study
Brief Title: Predictive Value of Postoperative Circulating Tumor DNA Monitoring for Colorectal Cancer Recurrence
Status: Active, not recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Collaborators: Guangzhou Burning Rock Dx Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Gong Chen, Professor, Sun Yat-sen University
Other Study IDs: pilotCRC-MRD
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Colorectal Cancer
Keywords: circulating tumor DNA; recurrence
MeSH Terms: conditions — Colorectal Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: Patients with stage I to IV colorectal cancer
  Interventions: Other: Serial ctDNA monitoring

INTERVENTIONS:
Other: Serial ctDNA monitoring — Baseline blood samples, surgical resected tumor tissue, blood samples after surgery (D5-7), blood samples before adjuvant therapy and blood samples after adjuvant therapy (every 3 months for up to 2 years follow-up) will be collected from colorectal patients.

SUMMARY:
This observational study aims to assess the predictive value of postoperative circulating tumor DNA (ctDNA) monitoring in evaluating the risk of recurrence in stage I-IV colorectal cancer patients. The study involves the collection of blood samples from patients who have undergone surgery for colorectal cancer. Sensitivity-enhanced molecular biology techniques are utilized to detect ctDNA in these samples. The correlation between ctDNA detection and the risk of recurrence is evaluated by analyzing patient follow-up data and clinical information. The findings of this study may contribute to the development of improved postoperative management strategies, such as identifying high-risk individuals and implementing additional treatment measures to reduce the risk of recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of signing the informed consent form.
2. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0-1.
3. Histologically confirmed colorectal cancer located from the ileocecal junction to the rectosigmoid junction, with a distance of >15cm from the anal verge. Regardless of mismatch repair (MMR) status, Rat sarcoma (RAS) gene and proto-oncogene serine/threonine-protein kinase (RAF) gene status.
4. Pathologically or cytologically confirmed American Joint Committee on Cancer (AJCC) tumor node metastasis (TNM) stage I-IV colorectal cancer patients (8th edition).
5. No evidence of distant metastasis confirmed by comprehensive examination (no distant organ or lymph node metastasis).
6. Normal organ function, as indicated by the following criteria:

   * Hematology criteria: For patients who have not received blood transfusion, white blood cell (WBC) ≥ 3.5/4.0 × 10^9/L, neutrophils ≥ 1.5 × 10^9/L, platelet (PLT) ≥ 100 × 10^9/L.
   * Biochemistry criteria: Crea and bilirubin (BIL) ≤ 1.0 times the upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times ULN, alkaline phosphatase (ALP) ≤ 2.5 × ULN, total bilirubin (Tbil) ≤ 1.5 × ULN.
7. Ability to provide clinical data required for the study.
8. Sufficient tumor tissue available for analysis.
9. Patients capable of achieving R0 radical resection.
10. Patients capable of adhering to the planned schedule, actively participating in regular clinical follow-up, and necessary treatments.

Exclusion Criteria:

1. History of concurrent or prior malignancies (excluding adequately treated cervical carcinoma in situ, basal cell carcinoma, or squamous cell carcinoma of the skin).
2. Patients who have received neoadjuvant therapy.
3. Patients with other severe diseases that may affect follow-up and short-term survival, as determined by the investigator.
4. Any other medical, social, or psychological conditions that, in the opinion of the investigator, would make the patient unsuitable for participation in this study.
5. Inability to undergo clinical follow-up using contrast-enhanced magnetic resonance imaging (MRI) or contrast-enhanced computed tomography (CT).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage I-IV colorectal cancer with curative intent.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
2-year recurrence free survival rate of the cohort evaluated by ctDNA | 2 years post surgery
  To evaluate the correlation between circulating tumor DNA (ctDNA) detection and recurrence-free survival.

SECONDARY OUTCOMES:
The ctDNA positive rate in stage III colorectal cancer | Within 4-6 week post operation
  To assess positive rate of ctDNA minimal residual disease (MRD) test in stage III of colorectal cancer patient after surgery.
Time point of ctDNA MRD test for recurrence monitoring | Within 4-6 week post operation
  To assess time from positive ctDNA test to clinical recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Gong Chen, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Siegel RL, Miller KD, Goding Sauer A, Fedewa SA, Butterly LF, Anderson JC, Cercek A, Smith RA, Jemal A. Colorectal cancer statistics, 2020. CA Cancer J Clin. 2020 May;70(3):145-164. doi: 10.3322/caac.21601. Epub 2020 Mar 5. PMID 32133645
- [Background] Govindarajan A, Fraser N, Cranford V, Wirtzfeld D, Gallinger S, Law CH, Smith AJ, Gagliardi AR. Predictors of multivisceral resection in patients with locally advanced colorectal cancer. Ann Surg Oncol. 2008 Jul;15(7):1923-30. doi: 10.1245/s10434-008-9930-1. Epub 2008 May 13. PMID 18473145
- [Background] Reinert T, Henriksen TV, Christensen E, Sharma S, Salari R, Sethi H, Knudsen M, Nordentoft I, Wu HT, Tin AS, Heilskov Rasmussen M, Vang S, Shchegrova S, Frydendahl Boll Johansen A, Srinivasan R, Assaf Z, Balcioglu M, Olson A, Dashner S, Hafez D, Navarro S, Goel S, Rabinowitz M, Billings P, Sigurjonsson S, Dyrskjot L, Swenerton R, Aleshin A, Laurberg S, Husted Madsen A, Kannerup AS, Stribolt K, Palmelund Krag S, Iversen LH, Gotschalck Sunesen K, Lin CJ, Zimmermann BG, Lindbjerg Andersen C. Analysis of Plasma Cell-Free DNA by Ultradeep Sequencing in Patients With Stages I to III Colorectal Cancer. JAMA Oncol. 2019 Aug 1;5(8):1124-1131. doi: 10.1001/jamaoncol.2019.0528. PMID 31070691
- [Derived] Cao D, Lv GZ, Li C, Wang FL, Zhou QX, Cai SL, Wu XJ, Jiang W, Yang X, Liu YF, Wu MQ, Li LR, Lu ZH, Pan ZZ, Lin JZ, Kong LH, Ding PR, Zhang DY, Yang JB, Lu SX, Peng JH, Mei WJ, Chen S, Sun Q, Chen SQ, Wan DS, Fan XN, Wang GQ, Li CC, Sun Y, Wu SL, Zhang ZH, Zhang RX, Chen G. Association of Recurrence with a Tumor-informed Personalized ctDNA Detection Approach in Resectable Colorectal Cancer: Results of a Prospective Observational Study. Ann Surg. 2025 Nov 3. doi: 10.1097/SLA.0000000000006971. Online ahead of print. PMID 41177967